CLINICAL TRIAL: NCT05422443
Title: The Turkish Adaptation, Validity, and Reliability Study of the Pain Coping Questionnaire
Brief Title: The Turkish Version of Pain Coping Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof. PhD, Akdeniz University
Other Study IDs: 2022-125
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
Keywords: pain; children; coping
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic pain group: Children with chronic pain
- Health group: children without chronic pain

SUMMARY:
Biological, psychological, and social factors all influence a child's sense of pain. Pain beliefs can have a significant impact on a person's perception of pain and adherence to treatment. As a result, pain management requires a thorough examination of the factors that influence pain perception. Coping is a cognitive and behavioral response to conditions and threats based on by personal or environmental factors. Children who do not have adequate coping mechanisms suffer from more severe pain. As a result, dealing with pain is a crucial part of pain management. This highlights the need of assessing pain coping in children when treating chronic pain. The purpose of this study is to show that the Turkish version of the Pain Coping Questionnaire (PCQ), which assesses children's pain coping techniques, is valid and reliable, as well as to ensure that it is culturally appropriate.

DETAILED DESCRIPTION:
Pain is a biopsychosocial term that comprises sensory, cognitive, and emotional factors. The biological, psychological, and cognitive aspects of pain are all present. Pain symptoms and comorbid symptoms are biological characteristics; anxiety, depression, and rage are psychological characteristics; and the ability to cope, catastrophize, and manage pain are cognitive characteristics. As a result, pain is influenced by a person's past experiences and beliefs. Pain that lasts longer than three months is referred to as chronic pain. A major issue is the high prevalence of chronic pain in children. Children with chronic pain have a lower quality of life than their healthy peers. Furthermore, this effect is unrelated to the degree of biological damage. Some children are more sensitive to pain than others, regardless of the severity of the condition. Because psychological, cognitive, and social variables influence an individual's perception of pain in addition to biological tissue damage.

The use of coping techniques in children varies based on the diagnosis, age, and gender of the child, according to the literature. Inadequate coping techniques are linked to a lower quality of life and increased pain severity. As a result, pain assessment in children with chronic pain should be done within a biopsychosocial framework. Various assessments have been developed to assess children's pain tolerating abilities. The Pain Coping Questionnaire (PCQ) was created to evaluate problem-focused, emotional-focused, and avoidance-focused coping strategies in children. It's the most commonly used scale for assessing children's coping techniques. The purpose of this study is to show that the Turkish version of the Pain Coping Questionnaire is valid and reliable (PCQ).

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 years and 18 years;
* Diagnosed with chronic pain.
* To have the cognitive ability to answer questions for assessment.
* Completing the test-retest assessment.
* To be able to read and speak Turkish

Exclusion Criteria:

* Patients with unmanageable psychological disorders (e.g., attention deficit hyperactivity disorder, autistic spectrum disorder, schizophrenia, bipolar disorder, major depressive disorder) would be excluded from the study.
* Patients who started a new treatment during the trial or 6 weeks before to the study for chronic pain.
* Those who take analgesics 48 hours prior to study evaluations

Inclusion Criteria for Healthy Children:

* Healthy children aged 6-18 years old
* Children without a psychiatric and neurological diagnosis

Exclusion Criteria for Healthy Children:

* Children got medical treatment for a neuropsychiatric disorder
* Children whose parents or themselves refused to participate

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children are diagnosed with chronic pain and their parents Children without chronic pain and their parents
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-08-08 (Estimated); Study Completion 2023-08-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of coping strategies | Baseline
  Pain Coping Questionnaire: Evaluates the coping strategies of children and adolescents with a total of 39 items in 8 subscale. These are seeking knowledge, problem solving, seeking social support, positive self-suggestion, behavioral distraction, cognitive distraction, externalization, and internalization/catastrophizing. Items are assessed on a 5-point Likert scale, with 1 indicating never and 5 indicating very often. Higher ratings indicate higher use of coping strategy. PCQ consists of parent and adolescent form.
Evaluation of pain | Baseline
  Wong baker faces pain scale: It is a valid and reliable scale preferred by children and their families to evaluate the severity of pain. It consists of 6 facial expressions that symbolize the severity of pain. These show the stages of increased pain from a smiling face (0 points) to a very sad and crying face (10 points). The meaning of each facial expression is carefully explained to the child. Children rate pain intensity according to face shapes.

SECONDARY OUTCOMES:
Evaluation of pain acceptance | Baseline
  Pain Flexibility Scale for Children: The scale assesses children's pain acceptance in chronic pain.It has a total of 20 questions divided into two sub-sections: valued activities and pain resistance. Pain resistance examines pain avoidance and control, whereas valued behaviors assesses involvement in meaningful activities despite pain. The scale is a seven-point Likert scale, with 0 indicating total disagreement (never true), and 6 indicating total agreement (Always true).

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, Assoc. Prof., Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study result will be published to the journal

REFERENCES:
- [Result] Liossi C, Howard RF. Pediatric Chronic Pain: Biopsychosocial Assessment and Formulation. Pediatrics. 2016 Nov;138(5):e20160331. doi: 10.1542/peds.2016-0331. Epub 2016 Oct 14. PMID 27940762
- [Result] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Result] Huguet A, Miro J. The severity of chronic pediatric pain: an epidemiological study. J Pain. 2008 Mar;9(3):226-36. doi: 10.1016/j.jpain.2007.10.015. Epub 2007 Dec 21. PMID 18088558
- [Result] Fraga MM, Terreri MT, Azevedo RT, Hilario MOE, Len CA. PAIN PERCEPTION AND PAIN COPING MECHANISMS IN CHILDREN AND ADOLESCENTS WITH JUVENILE FIBROMYALGIA AND POLYARTICULAR JUVENILE IDIOPATHIC ARTHRITIS. Rev Paul Pediatr. 2019 Jan-Mar;37(1):11-19. doi: 10.1590/1984-0462/;2019;37;1;00006. Epub 2018 Jun 11. PMID 29898009
- [Result] Failo A, Beals-Erickson SE, Venuti P. Coping strategies and emotional well-being in children with disease-related pain. J Child Health Care. 2018 Mar;22(1):84-96. doi: 10.1177/1367493517749326. Epub 2017 Dec 19. PMID 29258354
- [Result] Hermann C, Hohmeister J, Zohsel K, Ebinger F, Flor H. The assessment of pain coping and pain-related cognitions in children and adolescents: current methods and further development. J Pain. 2007 Oct;8(10):802-13. doi: 10.1016/j.jpain.2007.05.010. Epub 2007 Jul 12. PMID 17631054